CLINICAL TRIAL: NCT01567761
Title: A Prospective, Randomized and Double Blind Study on The Effect of Two Different Artificial Respiration Methods on the Intraocular Pressure During Surgery Under General Anesthesia
Brief Title: The Effect of Two Different Artificial Respiration Methods on the Intraocular Pressure During Surgery Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3111
Record Dates: First submitted 2012-03-29; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Intra Ocular Hypertension
Keywords: IOP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine whether the intraocular pressure of operated people under general anesthesia is affected by the artificial respiration method. If it is proven that there is such influence, the findings may lead to select the best method for patients with increased intraocular pressure.

In this study, the investigators will monitor the changes observed in intraocular pressure caused during an operation in two different artificial respiration methods:

1. Intermittent positive pressure ventilation (IPPV)
2. High frequency jet ventilation (HFJV)

Study recruited 50 patients aged 18 - 40, candidates to elective orthopedic surgery in the limbs. These patients do not suffer from general diseases that restrict their daily functioning.

The selection of the type of surgery was done to prevent the involvement of any other factor, except the respiration method, determination of intraocular pressure.

Exclusion Criteria:

* Patients who are unable to provide an Informed Consent
* Patients suffering from any eye disease
* Patients with corneal thickness less than 450 microns or more than 600 microns
* Smokers
* Patients with pulmonary disease restrictive or obstructive
* Patients using bronchodilator

All patients operated under general anesthesia using total intravenous anesthesia )TIVA) method.

All patients will be resuscitating half of the time of surgery using IPPV, and in the second half of surgery using HFJV.

During the surgery the IOP will be measured by an ophthalmologist who is unaware of the respiration method.

Correction will be made to the intraocular pressure values, depending on the thickness of the cornea.

The results of the measurements will be collected and the clinical significance will be reviewed by acceptable statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 40
* Patients candidates to elective orthopedic surgery in the limbs
* Patients do not suffer from general diseases that restrict their daily functioning.

Exclusion Criteria:

* Patients who are unable to provide an Informed Consent
* Patients suffering from any eye disease
* Patients with corneal thickness less than 450 microns or more than 600 microns
* Smokers
* Patients with pulmonary disease restrictive or obstructive
* Patients using bronchodilator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 18 - 40, candidates to elective orthopedic surgery in the limbs. These patients do not suffer from general diseases that restrict their daily functioning.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-05